CLINICAL TRIAL: NCT03968822
Title: The Use of Intralipid® 20% Solution to Reverse the Anesthetic Effect of Local Anesthetics: a Proof of Concept Study in Volunteers
Brief Title: Intralipid® 20% for Reversal of Local Anesthetics
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2018-2039
Record Dates: First submitted 2019-05-21; First posted 2019-05-30 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Anesthesia, Local
MeSH Terms: interventions — Lidocaine; Lidoderm; Bupivacaine; soybean oil, phospholipid emulsion; Salts; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be blinded to which treatment they are receiving both times they come in for the study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intralipid 20% IV Bolus (Experimental): This is 1 out of the 2 study visits. The patient will receive 6 injections (3 in each thigh). The 6 injections are:
  1. lidocaine 1%
  2. lidocaine 2%
  3. bupivacaine 0.5%
  4. bupivacaine 0.25%
  5. saline
  6. no injection
  Each test solution will be injected over 5 seconds through a 27G needle and tuberculin syringe at a 30 degree angle.
  The patient will also receive an intravenous bolus in the arm of Intralipid 20%.
  Participant will be blindfolded for these activities so they will not know what they received during the visit.
  Interventions: Drug: Lidocaine 2%; Drug: Lidocaine 1%; Drug: Bupivacaine 0.25%; Drug: Bupivacaine 0.5%; Drug: Intralipid, 20% Intravenous; Other: Saline
- Saline (Placebo Comparator): This is 2 out of the 2 study visits. The patient will receive 6 injections (3 in each thigh). The 6 injections are:
  1. lidocaine 1%
  2. lidocaine 2%
  3. bupivacaine 0.5%
  4. bupivacaine 0.25%
  5. saline
  6. no injection
  Each test solution will be injected over 5 seconds through a 27G needle and tuberculin syringe at a 30 degree angle.
  The patient will also receive an intravenous bolus in the arm of Saline.
  Participant will be blindfolded for these activities so they will not know what they received during the visit.
  Interventions: Drug: Lidocaine 2%; Drug: Lidocaine 1%; Drug: Bupivacaine 0.25%; Drug: Bupivacaine 0.5%; Other: Saline intravenously; Other: Saline

INTERVENTIONS:
Drug: Lidocaine 2% — 3 mL of test solution to a skin area on the thigh, 2cm in diameter
  Other Names: Lidocaine Viscous; Lidoderm; Recticare
Drug: Lidocaine 1% — 3 mL of test solution to a skin area on the thigh, 2cm in diameter
  Other Names: Lidocaine Viscous; Lidoderm; Recticare
Drug: Bupivacaine 0.25% — 3 mL of test solution to a skin area on the thigh, 2cm in diameter
  Other Names: Marcaine; Sensorcaine
Drug: Bupivacaine 0.5% — 3 mL of test solution to a skin area on the thigh, 2cm in diameter
  Other Names: Marcaine; Sensorcaine
Drug: Intralipid, 20% Intravenous — a 250ml bag administered intravenously
  Other Names: i.v. fat emulsion
  Arms: Intralipid 20% IV Bolus
Other: Saline intravenously — a 250ml bag administered intravenously
  Other Names: salt
  Arms: Saline
Other: Saline — 3 mL of test solution to a skin area on the thigh, 2cm in diameter
  Other Names: salt

SUMMARY:
In order to determine if Intralipid 20% can be used to reverse the effects of local anesthetics, the investigators will recruit 18 volunteers who will be asked to come to HSS for two study visits. Small amounts of local anesthetics will be injected into the volunteers' thighs during both visits. During one visit volunteers will receive Intralipid 20% and during the other visit they will receive a saline solution. The study team will measure how quickly normal sensation returns to the thighs when the volunteers get Intralipid 20% compared to saline.

DETAILED DESCRIPTION:
The purpose of this study is to determine if a fat solution (Intralipid 20%) given intravenously can reverse the effects of local anesthetics. Local anesthetics are drugs that cause numbness when they are injected into different parts of the body. Local anesthetics are important drugs because they allow doctors to perform surgeries and other procedures on patients; however, there are certain instances where it would be helpful to reverse the effects of local anesthetics and reduce the amount of time that they produce numbness. In order to determine if Intralipid 20% can be used to reverse the effects of local anesthetics, the investigators will recruit 18 volunteers who will be asked to come to HSS for two study visits. Small amounts of local anesthetics will be injected into the volunteers' thighs during both visits. During one visit volunteers will receive Intralipid 20% and during the other visit they will receive a saline solution. The study team will measure how quickly normal sensation returns to the thighs when the volunteers get Intralipid 20% compared to saline.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* BMI 18-25, with body weight between 50-100kg

Exclusion Criteria:

* ASA III or higher
* Pregnant Women
* Allergy to study medications (lidocaine, bupivacaine, soybeans, eggs)
* Use of drugs affecting the sensorium (including opioids, benzodiazepines, antipsychotics, gabapentinoids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-07-26 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Time to complete normal sensation after lidocaine 1% | up to 24 hours
  The time (measured in minutes) when the participant reports normal sensation of both cold swab and pinprick at the injection site of lidocaine 1%.
  Although measured for each individual participant, the average time across all participants is reported.
Time to complete normal sensation after lidocaine 2% | up to 24 hours
  The time (measured in minutes) when the participant reports normal sensation of both cold swab and pinprick at the injection site of lidocaine 2%.
  Although measured for each individual participant, the average time across all participants is reported.
Time to complete normal sensation after Bupivacaine 0.5% | up to 24 hours
  The time (measured in minutes) when the participant reports normal sensation of both cold swab and pinprick at the injection site of Bupivacaine 0.5%.
  Although measured for each individual participant, the average time across all participants is reported.
Time to complete normal sensation after Bupivacaine 0.25% | up to 24 hours
  The time (measured in minutes) when the participant reports normal sensation of both cold swab and pinprick at the injection site of Bupivacaine 0.25%.
  Although measured for each individual participant, the average time across all participants is reported.

SECONDARY OUTCOMES:
Time to normal cold swab sensation after lidocaine 1% | up to 24 hours
  The time (measured in minutes) when the participant reports normal sensation of cold swab at the injection site of lidocaine 1%.
  Although measured for each individual participant, the average time across all participants is reported.
Time to normal pinprick sensation after lidocaine 1% | up to 24 hours
  The time (measured in minutes) when the participant reports normal sensation of pinprick at the injection site of lidocaine 1%.
  Although measured for each individual participant, the average time across all participants is reported.
Time to normal cold swab sensation after lidocaine 2% | up to 24 hours
  The time (measured in minutes) when the participant reports normal sensation of cold swab at the injection site of lidocaine 2%.
  Although measured for each individual participant, the average time across all participants is reported.
Time to normal pin prick sensation after lidocaine 2% | up to 24 hours
  The time (measured in minutes) when the participant reports normal sensation of pinprick at the injection site of lidocaine 2%.
  Although measured for each individual participant, the average time across all participants is reported.
Time to normal pinprick sensation after Bupivacaine 0.5% | up to 24 hours
  The time (measured in minutes) when the participant reports normal sensation of pinprick at the injection site of Bupivacaine 0.5%.
  Although measured for each individual participant, the average time across all participants is reported.
Time to normal cold swab sensation after Bupivacaine 0.5% | up to 24 hours
  The time (measured in minutes) when the participant reports normal sensation of cold swab at the injection site of Bupivacaine 0.5%.
  Although measured for each individual participant, the average time across all participants is reported.
Time to normal cold swab sensation after Bupivacaine 0.25% | up to 24 hours
  The time (measured in minutes) when the participant reports normal sensation of cold swab at the injection site of Bupivacaine 0.25%.
  Although measured for each individual participant, the average time across all participants is reported.
Time to normal pinprick sensation after Bupivacaine 0.25% | up to 24 hours
  The time (measured in minutes) when the participant reports normal sensation of pinprick at the injection site of Bupivacaine 0.25%.
  Although measured for each individual participant, the average time across all participants is reported.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Memtsoudis, MD/PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital of Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures)
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. For individual participant meta-analysis. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our data warehouse but without investigator support other than deposited metadata.